CLINICAL TRIAL: NCT01755286
Title: A Prospective, Randomized, Double-Blind, Placebo- and Sham-Controlled, Multicenter, Phase 1b Study of OTO-201 Given as a Single Intratympanic Injection for Intra-Operative Treatment of Middle Ear Effusion in Pediatric Subjects Requiring Tympanostomy Tube Placement
Brief Title: OTO-201 for Middle Ear Effusion in Pediatric Subjects Requiring Tympanostomy Tube Placement
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otonomy, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 201-201101
Record Dates: First submitted 2012-12-18; First posted 2012-12-24 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Bilateral Middle Ear Effusion Requiring Tympanostomy Tube Placement
MeSH Terms: interventions — Ciprofloxacin; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 4 mg OTO-201 (Experimental)
  Interventions: Drug: OTO-201
- 12 mg OTO-201 (Experimental)
  Interventions: Drug: OTO-201
- Vehicle for OTO-201 (Placebo Comparator)
  Interventions: Drug: Placebo
- Sham (Sham Comparator)
  Interventions: Drug: Sham

INTERVENTIONS:
Drug: OTO-201 — Single intra-operative injection
  Other Names: ciprofloxacin
  Arms: 12 mg OTO-201; 4 mg OTO-201
Drug: Placebo — Single intratympanic injection
  Arms: Vehicle for OTO-201
Drug: Sham — Simulated single intratympanic injection
  Arms: Sham

SUMMARY:
The purpose of this study is to describe the safety and tolerability of two dose levels of OTO-201, placebo and sham when administered intra-operatively in pediatric subjects with bilateral middle ear effusion who require tympanostomy tube placement.

ELIGIBILITY:
Inclusion Criteria includes, but is not limited to:

* Subject is a male or female aged 6 months to 12 years, inclusive
* Subject has a clinical diagnosis of bilateral middle ear effusion requiring tympanostomy tube placement
* Subject's caregiver is willing to comply with the protocol and attend all study visits

Exclusion Criteria includes, but is not limited to:

* Subject has a history of prior ear or mastoid surgery, not including myringotomy or myringotomy with tympanostomy tube placement
* Subject has a history of sensorineural hearing loss
* Subject has a history of chronic or recurrent bacterial infections other than otitis media that likely will require treatment with antibiotics during the course of the study

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 83 (Actual)
Dates: Start 2012-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Safety | Up to 1 month
  Evaluation of adverse events, otoscopic exams, audiometry, and tympanometry

SECONDARY OUTCOMES:
Clinical Activity | Up to 1 month
  Evaluation of physician reported and caregiver reported otorrhea
Microbiological Eradication | Up to 1 month
  Microbiological eradication of pretherapy bacteria

CONTACTS AND LOCATIONS:
Overall Officials: Carl LeBel, PhD, Study Chair — Otonomy, Inc.
Locations (1):
- Call/Email Otonomy Central Contact for Trial Locations, San Diego, California, United States